CLINICAL TRIAL: NCT00591149
Title: Phase II Trial Of Oxaliplatin With Docetaxel Followed By Epidermal Growth Factor Antibody (EGFR-AB) Cetuximab In Patients With Recurrent Or Metastatic Squamous Cell Carcinoma of Head and Neck (SCCHN)
Brief Title: Oxaliplatin and Docetaxel Followed by Cetuximab for Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to termination of funding
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10635
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer; Carcinoma, Squamous
Keywords: cancer; head and neck cancer; squamous cell cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Neoplasms; Neoplasms, Squamous Cell | interventions — Oxaliplatin; Docetaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients will be treated with oxaliplatin 130 MG/M2 IV over 2 hours on day 1 and docetaxel 60 MG/M2 IV over 1 hour on day 1 of a 21 day cycle. Cycles of treatment will be repeated every 3 weeks for a total of 4 cycles or until disease progression or intolerable toxicity.
  Patients who were treated with 4 cycles of oxaliplatin and docetaxel and had a response or stable disease will be treated with cetuximab at 400 MG/M2 on week 1 then 250 MG/M2 weekly for a total of 12 weeks, or until disease progression or intolerable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: Docetaxel; Drug: Cetuximab

INTERVENTIONS:
Drug: Oxaliplatin — 130 MG/M2 IV over 2 hours on day 1 of 21 day cycle over a period of 4 cycles
  Other Names: Eloxatin
Drug: Docetaxel — 60 MG/M2 IV over 1 hour on day 1 of a 21 day cycle for a period of 4 cycles
  Other Names: Taxotere
Drug: Cetuximab — 400 MG/M2 on week 1 then 250 MG/M2 weekly for a total of 12 weeks
  Other Names: Erbitux

SUMMARY:
A study of Oxaliplatin and Docetaxel followed by Cetuximab for head and neck cancer patients to determine their effect on the control and reduction of tumor size

DETAILED DESCRIPTION:
This is a non-randomized, open-label, phase II study to assess the effects of oxaliplatin and docetaxel followed by epidermal factor-antibody (EGFR-AB) cetuximab on patients with previously treated recurrent /metastatic squamous cell carcinoma of the head and neck. Head and neck tissue will also be tested to determine if the protein Epidermal Growth Factor Receptor is present in the cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent SCCHN
* 18 years or older
* Tumor site accessible by biopsy
* Measurable disease
* Receiving no other therapy
* ECOG performance status 0-1
* Adequate bone marrow, renal function and hepatic function

Exclusion Criteria:

* Active infection or fever within 3 days of treatment
* Active CNS metastases
* Prior malignancy within 5 years
* Hypersensitivity to study drugs
* Chemotherapy within 30 days of treatment
* Concurrent investigational therapy within 30 days
* Radiotherapy of more than 25% of bone marrow
* Peripheral neuropathy of grade 2 or greater
* Pregnant or lactating patients
* History of allogeneic transplant
* Active or previously treated HIV or Hepatitis B or C
* Patients with a tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chao Huang, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxaliplatin and Docetaxel: Patients will be treated with oxaliplatin 130 MG/M2 IV over 2 hours on day 1 and docetaxel 60 MG/M2 IV over 1 hour on day 1 of a 21 day cycle. Cycles of treatment will be repeated every 3 weeks for a total of 4 cycles or until disease progression or intolerable toxicity.
  Patients who were treated with 4 cycles of oxaliplatin and docetaxel and had a response or stable disease will be treated with cetuximab at 400 MG/M2 on week 1 then 250 MG/M2 weekly for a total of 12 weeks, or until disease progression or intolerable toxicity.
  Docetaxel : 60 MG/M2 IV over 1 hour on day 1 of a 21 day cycle for a period of 4 cycles
  Cetuximab : 400 MG/M2 on week 1 then 250 MG/M2 weekly for a total of 12 weeks
  Oxaliplatin : 130 MG/M2 IV over 2 hours on day 1 of 21 day cycle over a period of 4 cycles
Period: Overall Study
Arm/Group | Oxaliplatin and Docetaxel
Started | 16
Completed | 11
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Oxalipatin and Docetaxel: Patients will be treated with oxaliplatin 130 MG/M2 IV over 2 hours on day 1 and docetaxel 60 MG/M2 IV over 1 hour on day 1 of a 21 day cycle. Cycles of treatment will be repeated every 3 weeks for a total of 4 cycles or until disease progression or intolerable toxicity.
  Patients who were treated with 4 cycles of oxaliplatin and docetaxel and had a response or stable disease will be treated with cetuximab at 400 MG/M2 on week 1 then 250 MG/M2 weekly for a total of 12 weeks, or until disease progression or intolerable toxicity.
  Oxaliplatin: 130 MG/M2 IV over 2 hours on day 1 of 21 day cycle over a period of 4 cycles
  Docetaxel: 60 MG/M2 IV over 1 hour on day 1 of a 21 day cycle for a period of 4 cycles
  Cetuximab: 400 MG/M2 on week 1 then 250 MG/M2 weekly for a total of 12 weeks
Arm/Group | Oxalipatin and Docetaxel
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 66 [51 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Measured by Response Rate in Participants
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT and MRI:
  * Complete Response (CR), Disappearance of all target lesions;
  * Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions;
  * Stable Disease (NR/SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since the treatment started;
  * Progressive Disease (PD), A 20% or greater increase in the sum of the longest diameter of measured lesions (target lesions), taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 12 Weeks, 1 Year
Measure: Number; unit: participants
Groups:
- Oxaliplatin and Docetaxel: Patients will be treated with oxaliplatin 130 MG/M2 IV over 2 hours on day 1 and docetaxel 60 MG/M2 IV over 1 hour on day 1 of a 21 day cycle. Cycles of treatment will be repeated every 3 weeks for a total of 4 cycles or until disease progression or intolerable toxicity.
  Patients who were treated with 4 cycles of oxaliplatin and docetaxel and had a response or stable disease will be treated with cetuximab at 400 MG/M2 on week 1 then 250 MG/M2 weekly for a total of 12 weeks, or until disease progression or intolerable toxicity.
  Oxaliplatin: 130 MG/M2 IV over 2 hours on day 1 of 21 day cycle over a period of 4 cycles
  Docetaxel: 60 MG/M2 IV over 1 hour on day 1 of a 21 day cycle for a period of 4 cycles
  Cetuximab: 400 MG/M2 on week 1 then 250 MG/M2 weekly for a total of 12 weeks
Arm/Group | Oxaliplatin and Docetaxel
Number analyzed (Participants) | 16
participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 6
  Progressive Disease | 3
  Not Evaluable | 5

ADVERSE EVENTS:
Arm/Group | Oxaliplatin and Docetaxel
Serious Adverse Events (participants affected / at risk) | 10/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin and Docetaxel (N=16)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Infection, lung (Pneumonia) (Infections and infestations) | 2 (3)
Multi-organ failure (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin and Docetaxel (N=16)
Alanine aminotrasferase increased (Investigations) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (6)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (8)
Aspartate aminotrasferase increased (Investigations) | 4 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Bruising (Injury, poisoning and procedural complications) | 1 (3)
Colitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Creatinine increased (Investigations) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Abnormal ear, nose and throat examination (Ear and labyrinth disorders) | 1 (1)
Edema: limbs (General disorders) | 2 (2)
Edema: Head and Neck (General disorders) | 1 (1)
Elevated Alkaline Phosphatase (Investigations) | 1 (1)
Elevated blood urea nitrogen (Investigations) | 2 (3)
Esophagitis (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 10 (20)
Fever (Infections and infestations) | 3 (5)
Gastritis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hearing (Ear and labyrinth disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 2 (4)
Hemolysis (Blood and lymphatic system disorders) | 5 (12)
Hiccup (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 5 (17)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 5 (11)
Infection, mucosa (Infections and infestations) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 9 (21)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness: lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7)
Tissue necrosis: neck (Skin and subcutaneous tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (13)
Decreased platelets (Blood and lymphatic system disorders) | 5 (7)
Lung infection: Pneumonia (Infections and infestations) | 2 (2)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (6)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
dysgeusia (Nervous system disorders) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes